CLINICAL TRIAL: NCT03325660
Title: The Role of Whole Body Vibration and Pelvic Floor Muscle Exercises in Treating Urinary Incontinence Following Prostate Cancer Surgery: A Comparative Randomized Controlled Trial
Brief Title: Whole Body Vibration and Pelvic Floor Exercises on Urinary Incontinence
Acronym: [PTREC]
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahlia University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Dr Sayed Tantawy, Associate Professor, Ahlia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T. REC/012/001250
Record Dates: First submitted 2017-10-26; First posted 2017-10-30 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Urinary Incontinence
Keywords: Whole body vibration, Pelvic floor muscle
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The study group included 30 patients participated in pelvic floor muscle training and whole-body vibrations, 3 times weekly for 4 consecutive weeks; the frequency and peak-to-peak displacement of vibration were 2 mm/20 Hz for the first week for 5 minutes, 3mm/25 Hz, 10 minutes for the second week and 4 mm/30 Hz, 15 minutes for the last two weeks. The control group included 31 patients received only pelvic floor training only. Pelvic floor exercises: Each patient was prepared and taught a program of pelvic floor exercises to be performed in daily sessions in lying, sitting, and standing positions consisting of 10 seconds of contractions followed by 10 seconds of relaxation and repeating the exercises 15 times each session.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- study group (Active Comparator): whole body vibration
  Interventions: Other: whole body vibration
- control group (No Intervention): No intervention

INTERVENTIONS:
Other: whole body vibration — pelvic floor exercises
  Other Names: pelvic floor exercises
  Arms: study group

SUMMARY:
Stress urinary incontinence is common in men following prostate cancer surgery. Rehabilitative interventions incorporate pelvic floor muscle training, biofeedback, electrical stimulation, lifestyle changes, or a combination of these strategies. However, little is known about the physiological impact of whole-body vibration for stress urinary incontinence following radical prostatectomy. Participants: Sixty-one patients with mild Stress urinary incontinence after radical prostatectomy.

Intervention: patients were randomly assigned into two groups: group 1 included 30 patients who received pelvic floor muscle training and whole-body vibration training with a frequency and amplitude of 20 Hz/ 2 mm for the first 2 sessions and 40 Hz/ 4 mm for the rest of intervention; while group 2 included 31 patients who performed only pelvic floor muscle training. The intervention in both groups was performed three times per week for 4 weeks.

DETAILED DESCRIPTION:
Participants were recruited from Cairo University Hospitals who suffered from mild SUI for at least 6 months after RP. The diagnosis was confirmed by the referred physician via 24-h pad test which supposed to be less than 100 grams gain of weight of the pad/s worn by the patient.

The exclusion criteria were artificial pacemaker, body mass index (BMI)> 35 kg/m2, urinary infection, bleeding from the urinary bladder or the digestive tract, polyuria, diabetes mellitus, detrusor over-activity, neuromuscular disorder, ear problems or any other medical condition that would affect participation in the training program. Main outcomes: Incontinence Visual Analogue Scale (I-VAS), the International Consultation on Incontinence Questionnaire-Urinary Incontinence-Short Form (ICIQ-UI-SF) and 24-hour pad test.

ELIGIBILITY:
Inclusion Criteria:

* The initial sample was adult patients suffering from urinary incontinence at least 6 months after radical prostatectomy.

Exclusion Criteria:

* The exclusion criteria included patients with an artificial pacemaker, body mass index more than 35 kg/ m2, urinary infection, bleeding from the urinary bladder or the digestive tract, polyuria, diabetes mellitus, detrusor instability, neuromuscular disorders, and any other medical condition that affects participation in the training program.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — male patients suffering from urinary incontinence after prostate cancer surgery
Enrollment: 61 (Actual)
Dates: Start 2016-07-03 (Actual); Primary Completion 2017-03-05 (Actual); Study Completion 2017-10-27 (Actual)

PRIMARY OUTCOMES:
Incontinence Visual Analogue Scale (I-VAS) | 7 months
  For the I-VAS, patients were asked to depict their subjective burden of incontinence on a 100-mm VAS. The question above the VAS line was: 'How annoyed are you by incontinence currently?' The 100-mmVAS scale scores ranged from 0 ('not irritated') to 10 ('extremely disturbed'). A 100-mm line labelled from 0 to 10 was used, with patients asked to mark their answer on the line. The I-VAS is a valid, reproducible and responsive tool for UI treatment and improving the quality of life of patients after urogynaecologic surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sayed A A Tantawy, PhD, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tantawy SA, Elgohary HMI, Abdelbasset WK, Kamel DM. Effect of 4 weeks of whole-body vibration training in treating stress urinary incontinence after prostate cancer surgery: a randomised controlled trial. Physiotherapy. 2019 Sep;105(3):338-345. doi: 10.1016/j.physio.2018.07.013. Epub 2018 Sep 25. PMID 30630622